CLINICAL TRIAL: NCT05401071
Title: Efficacy and Safety of Short-course Treatment for Drug-sensitive Tuberculosis in China
Brief Title: Optimizing(O) RIfapentine-based(RI) Regimen and shortENing(EN) the Treatment of Drug-sensitive Tuberculosis(T)
Acronym: ORIENT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORIENT
Record Dates: First submitted 2022-02-27; First posted 2022-06-02 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis, Pulmonary
Keywords: rifapentine; shorter treatment; pulmonary tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Short Regimen with Rifapentine 10mg/kg (Experimental): Intervention: Short Regimen with Rifapentine 10mg/kg consists of two periods of 17- 26 weeks. The first is an intensive phase of 8 weeks, and included rifapentine, isoniazid, pyrazinamide, and moxifloxacin. This is followed by a continuation phase of 9 weeks with the following agents: rifapentine, isoniazid and moxifloxacin (extended up a maximum of 18 weeks if no smear conversion at the end of 8 weeks or the tuberculosis cavity is not closed at the end of 17 weeks).
  Interventions: Other: Short Regimen with Rifapentine 10mg/kg
- Short Regimen with Rifapentine 15mg/kg (Experimental): Intervention: Short Regimen with Rifapentine 15mg/kg consists of two periods of 17- 26 weeks. The first is an intensive phase of 8 weeks, and included rifapentine, isoniazid, pyrazinamide, and moxifloxacin. This is followed by a continuation phase of 9 weeks with the following agents: rifapentine, isoniazid and moxifloxacin (extended up a maximum of 18 weeks if no smear conversion at the end of 8 weeks or the tuberculosis cavity is not closed at the end of 17 weeks).
  Interventions: Other: Short Regimen with Rifapentine 15mg/kg
- Standardized Regimen (Active Comparator): Intervention：World Health Organization (WHO) Standardized Regimen group consists of 26 weeks with two phases of treatment. The first is an intensive phase of 8 weeks, and included rifampicin, isoniazid, pyrazinamide, and ethambutol. This is followed by a continuation phase of 18 weeks with the following agents: rifampicin and isoniazid.
  Interventions: Combination Product: Standardized Regimen
- Short Regimen with Rifapentine 20mg/kg (Experimental): Intervention: Short Regimen with Rifapentine 20mg/kg consists of two periods of 17- 26 weeks. The first is an intensive phase of 8 weeks, and included rifapentine, isoniazid, pyrazinamide, and moxifloxacin. This is followed by a continuation phase of 9 weeks with the following agents: rifapentine, isoniazid and moxifloxacin (extended up a maximum of 18 weeks if no smear conversion at the end of 8 weeks or the tuberculosis cavity is not closed at the end of 17 weeks).
  Interventions: Other: Short Regimen with Rifapentine 20mg/kg

INTERVENTIONS:
Other: Short Regimen with Rifapentine 10mg/kg — rifapentine 10mg/kg daily; isoniazid 300mg daily; pyrazinamide ≤50kg 1000mg daily, 50-71kg 1200mg daily, >71kg 1000mg daily; moxifloxacin 400mg daily. All treatment is taken orally.
  Arms: Short Regimen with Rifapentine 10mg/kg
Combination Product: Standardized Regimen — During the intensive phase, rifampicin ≤55kg 450mg daily, 55-71kg 600mg daily, >71kg 750mg daily; isoniazid ≤55kg 225mg daily, 55-71kg 300mg daily, >71kg 375mg daily; pyrazinamide ≤55kg 900mg daily, 55-71kg 1200mg daily, >71kg 1600mg daily; ethambutol ≤55kg 825mg daily, 55-71kg 1100mg daily, >71kg 1375mg daily; All treatment is taken orally.
  During the continuation phase, rifampicin ≤50kg 450mg daily, >50kg 600mg daily; isoniazid 300mg daily; All treatment is taken orally.
  Arms: Standardized Regimen
Other: Short Regimen with Rifapentine 15mg/kg — rifapentine 15mg/kg daily; isoniazid 300mg daily; pyrazinamide ≤50kg 1000mg daily, 50-71kg 1200mg daily, >71kg 1000mg daily; moxifloxacin 400mg daily. All treatment is taken orally.
  Arms: Short Regimen with Rifapentine 15mg/kg
Other: Short Regimen with Rifapentine 20mg/kg — rifapentine 20mg/kg daily; isoniazid 300mg daily; pyrazinamide ≤50kg 1000mg daily, 50-71kg 1200mg daily, >71kg 1000mg daily; moxifloxacin 400mg daily. All treatment is taken orally.
  Arms: Short Regimen with Rifapentine 20mg/kg

SUMMARY:
Tuberculosis (TB) remains the most important infectious disease in the world. A major barrier to tuberculosis control is poor adherence to long-term and complex treatment regimens.

This is a multicenter prospective, non-inferiority randomized controlled study. The purpose of our study is a) to evaluate the tolerability, efficacy and pharmacokinetics/pharmacodynamics (PK/PD) of the high-dose rifapentine, b) to evaluate whether the high-dose rifapentine-containing regimen has the potential to treat the rifampicin-sensitive pulmonary tuberculosis and shorten the course of treatment to 17 weeks. This study is of great significance for shortening the course of treatment, reducing the adverse reactions and economic burden of patients' treatment in rifampicin-sensitive tuberculosis patient.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the most important infectious disease in the world. A major barrier to tuberculosis control is poor adherence to long-term and complex treatment regimens. Incomplete TB treatment can lead to increased morbidity and mortality, prolonged infectivity and transmission, and the development of drug resistance. The development of new therapeutic strategies with stronger bactericidal activity could lead to shorter and better-tolerated regimens, thereby increasing cure rates, lowering costs, potentially reducing transmission and preventing the emergence of multidrug-resistant tuberculosis (MDR-TB).

This trial is a multicenter prospective, non-inferiority randomized controlled study. Rifampicin-sensitive pulmonary tuberculosis patients will be included in our study. Stage 1 of the study is designed to evaluate the tolerability, efficacy and PK/PD of the high-dose rifapentine in order to select two doses to carry forward into study Stage 2. Study Stage 2 will provide pivotal confirmation of efficacy, safety, and tolerability of the selected rifapentine doses in patients with rifampicin-sensitive pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years;
* Weight between 40 to 80 kg;
* Individuals with smear-positive pulmonary tuberculosis and sensitive to rifampicin ;
* Willing to provide signed informed consent, or parental consent and participant assent.
* If you are a non-menopausal woman, agree to use or have used effective contraception during treatment.

Exclusion Criteria:

* Combined extrapulmonary tuberculosis;
* Patients with extensive lesion (extent of disease greater than 50% or cavity size greater than 4cm) ;
* Individuals will be excluded from enrollment if, at the time of enrollment, their M. tuberculosis isolate is already known to be resistant to any one or more of the following: rifampin, isoniazid, pyrazinamide, ethambutol, or fluoroquinolones;
* Alcohol abuse#drinking more than 64g of ethanol a day for male, 42g for female#;
* Hemoglobin is less than 70g/L or platelet is less than 100*10^9/L;
* Patients with impaired liver function (hepatic encephalopathy, ascites; total bilirubin is higher than the upper limit of normal; Alanine aminotransferase or aspartate aminotransferase is higher than the upper limit of normal);
* Blood creatinine is more than 1.5 times the upper limit of normal;
* More than five days of systemic treatment with any one or more of the following drugs within 6 months preceding initiation of study drugs: isoniazid, rifampin, rifabutin, rifapentine, ethambutol, pyrazinamide, kanamycin, amikacin, streptomycin, capreomycin, moxifloxacin, levofloxacin, gatifloxacin, ofloxacin, ciprofloxacin, other fluoroquinolones, ethionamide, prothionamide, cycloserine, terizidone, para-aminosalicylic acid, linezolid, clofazimine, delamanid or bedaquiline;
* Known history of prolonged QT syndrome;
* Current or planned use within six months following enrollment of one or more of the following medications: HIV protease inhibitors, HIV integrase inhibitors, HIV entry and fusion inhibitors, HIV non-nucleoside reverse transcriptase inhibitors other than efavirenz; quinidine, procainamide, amiodarone, sotalol, disopyramide, ziprasidone, or terfenadine;
* Known allergy or intolerance to any of the study medications;
* AIDS patients;
* Pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2442 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate of the short regimen during drug treatment and follow-up. | 108 weeks after randomization
  To compare the treatment success rate without relapse between the short regimen with rifapentine 10mg/kg, the short regimen with rifapentine 15mg/kg, the short regimen with rifapentine 20mg/kg and the WHO standardized regimen group.

SECONDARY OUTCOMES:
The frequency of grade 3 or greater adverse events among patients Over the 108 Week Treatment and Follow-up Period. | up to 108 weeks
  To compare the proportion of patients who experience grade 3 or greater adverse events between the short regimen with rifapentine 10mg/kg, the short regimen with rifapentine 15mg/kg, the short regimen with rifapentine 20mg/kg and the WHO standardized regimen group.
Relapse rate during follow-up. | 82-91 weeks after the end of drug treatment.
  To compare the treatment success rate without relapse between the short regimen with rifapentine 10mg/kg, the short regimen with rifapentine 15mg/kg, the short regimen with rifapentine 20mg/kg and the WHO standardized regimen group.
the percentage of participants found to be culture-negative at the end of intensive phase and the end of treatment phase | 8 weeks, 17 weeks and 26 weeks after randomization
  To compare the percentage of participants found to be culture-negative at the end of intensive phase and the end of treatment phase between the short regimen with rifapentine 10mg/kg, the short regimen with rifapentine 15mg/kg, the short regimen with rifapentine 20mg/kg and the WHO standardized regimen group.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PhD., Principal Investigator — Huashan Hospital of Fudan University，Shanghai，China
Locations (6):
- China (6):
  - Guiyang Public Health Clinical Center, Guiyang, Guizhou
  - People's Hospital of Qiandongnan, Kaili, Guizhou
  - The Third People's Hospital of Liupanshui, Liupanshui, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Department of Infectious Disease, Huashan Hospital, Shanghai, Shanghai Municipality
  - People's Hospital of Zhuji, Zhejiang Province, Zhuji, Zhejiang

REFERENCES:
- [Derived] Feng Z, Miao Y, Peng Y, Sun F, Zhang Y, Li R, Ge S, Chen X, Song L, Li Y, Wang X, Zhang W. Optimizing (O) rifapentine-based (RI) regimen and shortening (EN) the treatment of drug-susceptible tuberculosis (T) (ORIENT) using an adaptive seamless design: study protocol of a multicenter randomized controlled trial. BMC Infect Dis. 2023 May 8;23(1):300. doi: 10.1186/s12879-023-08264-2. PMID 37158831